CLINICAL TRIAL: NCT04946136
Title: The Effect of Gait Modification on Knee Joint Load in Persons With Medial Tibiofemoral Osteoarthritis - A Pilot Study
Brief Title: Gait Modification and Knee Joint Load
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Awaiting additional funding
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Alison Chang, Associate Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00212048
Record Dates: First submitted 2021-06-15; First posted 2021-06-30 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Masking Description: This is a pilot single-arm study examining the effect of an intervention on biomechanical and symptomatic outcomes. There is no control group, therefore no masking employed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gait modification (Experimental): In this pilot study, participants modify their gait patterns guided by real-time visual feedback on their medial knee load while walking on an instrumented treadmill.
  Interventions: Other: Gait modification

INTERVENTIONS:
Other: Gait modification — Individualized gait modifications guided by real-time visual feedback of knee load

SUMMARY:
This pilot study aims to assess the effect of a 6-week individualized gait retraining program on knee load and symptoms in persons with knee osteoarthritis (OA).

DETAILED DESCRIPTION:
This study aims to pilot-test an individualized gait retraining intervention to reduce knee load, guided by real-time visual feedback of the external knee adduction moment (KAM), a commonly used determinant for medial tibiofemoral (TF) joint load, during walking. Our central hypothesis is that individuals with predominantly medial TF OA can adapt their gait patterns to lower KAM during walking; consequently, reduce knee load and pain.

ELIGIBILITY:
Inclusion Criteria:

* people with radiographic TF OA fulfilling American College of Rheumatology classification criteria
* reporting average knee pain on walking > 3 on an 11-point scale (0-10) in at least one knee
* pain or tenderness predominantly located on the medial knee.

Exclusion Criteria:

* medial TF joint space width greater than lateral
* Kellgren/Lawrence (K/L) grade 4
* knee surgery or intra-articular corticosteroid injection in the past 6 months
* uncomfortable walking on treadmill for 20 minutes
* unable to walk without a walking aide
* inflammatory arthritis
* other musculoskeletal or neurological disorders that affect gait patterns
* currently receiving physical therapy

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-01-11 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
External knee adduction moment during walking | Baseline-to-6-week change
  The external knee adduction moment during walking will be assessed using a10-camera optical motion capture system and force plates. A visual 3D program will be used to compute and plot the pre- and post-intervention external knee adduction moment during walking.
WOMAC (Western Ontario and McMaster Universities) score | Baseline-to-6-week change
  WOMAC questionnaire contains 24 questions in three domains of pain (score range 0-20), stiffness (score range 0-8) and physical function (score range 0-68). Higher score indicates worse symptom/function.

SECONDARY OUTCOMES:
External knee flexion moment during walking | Baseline-to-6-week change
  The external knee flexion moment during walking will be assessed using a10-camera optical motion capture system and force plates. A visual 3D program will be used to compute and plot the pre- and post-intervention external knee flexion moment during walking.
KOOS (Knee Injury and Osteoarthritis Outcome Score) | Baseline-to-6-week change
  KOOS questionnaire contains 42 items in 5 domains of pain, other symptoms, function in daily living, function in sport and recreation, and knee-related quality of life. Scores are transformed to a 0-100 scale, with 0 representing extreme knee problems and 100 representing no problems.

CONTACTS AND LOCATIONS:
Overall Officials: Alison H Chang, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States